CLINICAL TRIAL: NCT03871257
Title: A Phase 3 Randomized Study of Selumetinib Versus Carboplatin/Vincristine in Newly Diagnosed or Previously Untreated Neurofibromatosis Type 1 (NF1) Associated Low-Grade Glioma (LGG)
Brief Title: A Study of the Drugs Selumetinib Versus Carboplatin/Vincristine in Patients With Neurofibromatosis and Low-Grade Glioma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-01396; NCI-2019-01396 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACNS1831 (Other: Children's Oncology Group); ACNS1831 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2019-03-11; First posted 2019-03-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Low Grade Glioma; Neurofibromatosis Type 1; Visual Pathway Glioma
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Carboplatin; Magnetic Resonance Spectroscopy; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (carboplatin, vincristine) (Active Comparator): INDUCTION: Patients receive carboplatin IV over 60 minutes on days 1, 8, 15, 22, 43, 50, 57, and 64 and vincristine IV or IV push over 1 minute on days 1, 8, 15, 22, 29, 36, 43, 50, 57, and 64 in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI throughout the trial.
  MAINTENANCE: Patients receive carboplatin IV over 60 minutes on days 1, 8, 15, and 22 of each cycle and vincristine IV or IV push over 1 minute on days 1, 8, and 15 of each cycle. Cycles repeat every 6 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI throughout the trial.
  Interventions: Drug: Carboplatin; Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Vincristine Sulfate
- Arm II (selumetinib sulfate) (Experimental): Patients receive selumetinib sulfate PO BID on days 1-28 of each cycle. Treatment is continuous and cycles repeat every 28 days for 27 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI throughout the trial.
  Interventions: Procedure: Magnetic Resonance Imaging; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Selumetinib Sulfate

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm I (carboplatin, vincristine)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Selumetinib Sulfate — Given PO
  Other Names: AZD-6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulfate; AZD6244 Hydrogen Sulphate; Koselugo; Selumetinib Sulphate
  Arms: Arm II (selumetinib sulfate)
Drug: Vincristine Sulfate — Given IV or IV push
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Arm I (carboplatin, vincristine)

SUMMARY:
This phase III trial studies if selumetinib works just as well as the standard treatment with carboplatin/vincristine (CV) for subjects with NF1-associated low grade glioma (LGG), and to see if selumetinib is better than CV in improving vision in subjects with LGG of the optic pathway (vision nerves). Selumetinib is a drug that works by blocking some enzymes that low-grade glioma tumor cells need for their growth. This results in killing tumor cells. Chemotherapy drugs, such as carboplatin and vincristine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether selumetinib works better in treating patients with NF1-associated low-grade glioma compared to standard therapy with carboplatin and vincristine.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the efficacy of treatment with selumetinib sulfate (selumetinib) as measured by event-free survival (EFS) is non-inferior to treatment with carboplatin/vincristine sulfate (vincristine) (CV) in previously untreated neurofibromatosis type 1 (NF1)-associated low-grade glioma (LGG).

II. To determine whether visual acuity (VA) using Teller acuity cards (TAC), in patients with NF1-associated LGG within the optic pathway, is better in those treated with selumetinib compared to CV.

SECONDARY OBJECTIVES:

I. To estimate tumor response rates and overall survival (OS) in each treatment regimen in previously untreated NF1-associated LGG.

II. To evaluate VA outcomes utilizing HOTV letter acuity testing in previously untreated NF1-associated LGG within the optic pathway in patients who are old enough to perform visual acuity testing utilizing HOTV (a recognition acuity measure).

III. To describe the improvement in motor function as measured by the Vineland scale in patients with previously untreated NF1-associated LGG that have documented motor deficits at enrollment.

IV. To prospectively evaluate and compare the quality of life among patients treated with selumetinib or CV.

V. To prospectively evaluate and compare the cognitive, social, emotional, and behavioral functioning of patients with NF1-associated LGG treated with either selumetinib or CV.

EXPLORATORY OBJECTIVES:

I. To evaluate optical coherence tomography (OCT) measures of retinal axon and ganglion cell thickness as a marker of treatment response in previously untreated NF1-associated LGG within the optic pathway.

II. To compare novel, semi-automated volumetric magnetic resonance imaging (MRI) measures to traditional measurements of treatment response (bi-dimensional MRI measurements) in NF1-associated optic pathway tumors.

III. To obtain paired blood and tumor tissue to be banked for future NF1-LGG biology studies involving comprehensive molecular analysis, including but not limited to whole exome and ribonucleic acid (RNA) sequencing.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I:

INDUCTION: Patients receive carboplatin intravenously (IV) over 60 minutes on days 1, 8, 15, 22, 43, 50, 57, and 64 and vincristine IV on days 1, 8, 15, 22, 29, 36, 43, 50, 57, and 64 in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI throughout the trial.

MAINTENANCE: Patients receive carboplatin IV over 60 minutes on days 1, 8, 15, and 22 of each cycle and vincristine IV on days 1, 8, and 15 of each cycle. Cycles repeat every 6 weeks for 8 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI throughout the trial.

ARM II: Patients receive selumetinib sulfate orally (PO) twice daily (BID) on days 1-28 of each cycle. Treatment is continuous and cycles repeat every 28 days for 27 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo MRI throughout the trial.

After completion of study treatment, patients are followed up with MRIs and physical exams every 3 months for 1 year, every 6 months for 2 years, and then once yearly for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >= 2 years and =< 21 years at the time of enrollment
* Patients must have a body surface area (BSA) of >= 0.5 m^2 at enrollment
* Patients must have neurofibromatosis type 1 (NF1) based on clinical criteria and/or germline genetic testing
* Patients must be newly diagnosed or have previously diagnosed NF-1 associated LGG that has not been treated with any modality other than surgery
* For patients with optic pathway gliomas (OPGs):

  * Newly-diagnosed patients with OPG are eligible if there are neurologic symptoms (including visual dysfunction, as defined below) or other exam findings associated with the tumor
  * Previously-diagnosed patients with OPG are eligible if they have new or worsening neurologic symptoms (including visual dysfunction, as defined below) or have tumor growth
  * For both newly-diagnosed and previously-diagnosed OPG, the patient may be eligible, irrespective of whether there has been tumor growth or other neurological symptoms or worsening, if they meet at least one of the following visual criteria:

    * Visual worsening, defined as worsening of visual acuity (VA) or visual fields (VF) documented within the past year (by examination or history); OR
    * Significant visual dysfunction (defined as VA worse than normal for age by 0.6 logMAR [20/80, 6/24, or 2.5/10] or more in one or both eyes)
* For patients with LGG in other locations (i.e., not OPGs):

  * Newly-diagnosed patients with LGG are eligible if there are neurologic symptoms or other exam findings associated with the tumor

    * NOTE: Newly-diagnosed patients with LGG without associated neurologic symptoms or exam findings are not eligible
  * Previously-diagnosed patients with LGG are eligible if they have new or worsening neurologic symptoms or have tumor growth
* Although not required, if a biopsy/tumor resection is performed, eligible histologies will include all tumors considered LGG or low-grade astrocytoma (World Health Organization [WHO] grade I and II) by 5th edition WHO classification of central nervous system (CNS) tumors with the exception of subependymal giant cell astrocytoma
* Patients must have two-dimensional measurable tumor >= 1 cm^2
* Patients with metastatic disease or multiple independent primary LGGs are allowed on study
* Creatinine clearance or radioisotope glomerular filtration Rate (GFR) >= 70 mL/min/1.73 m^2 OR a serum creatinine based on age/sex (within 7 days prior to enrollment) as follows:

  * Age; maximum serum creatinine (mg/dL)
  * 2 to < 6 years; 0.8 (male) and 0.8 (female)
  * 6 to < 10 years; 1 (male) and 1 (female)
  * 10 to < 13 years; 1.2 (male) and 1.2 (female)
  * 13 to < 16 years; 1.5 (male) and 1.4 (female)
  * >= 16 years; 1.7 (male) and 1.4 (female)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age (within 7 days prior to enrollment) (children with a diagnosis of Gilbert's syndrome will be allowed on study regardless of their total and indirect [unconjugated] bilirubin levels as long as their direct [conjugated] bilirubin is < 3.1 mg/dL)
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 3 x upper limit of normal (ULN) = 135 U/L (within 7 days prior to enrollment). For the purpose of this study, the ULN for SGPT is 45 U/L
* Albumin >= 2 g/dL (within 7 days prior to enrollment)
* Left ventricular ejection fraction (LVEF) >= 53% (or institutional normal; if the LVEF result is given as a range of values, then the upper value of the range will be used) by echocardiogram (within 4 weeks prior to enrollment)
* Corrected QT (QTc) interval =< 450 msec by electrocardiography (EKG) (within 4 weeks prior to enrollment)
* Absolute neutrophil count >= 1,000/uL (unsupported) (within 7 days prior to enrollment)
* Platelets >= 100,000/uL (unsupported) (within 7 days prior to enrollment)
* Hemoglobin >= 8 g/dL (may be supported) (within 7 days prior to enrollment)
* Patients with a known seizure disorder should be stable and should have not experienced a significant increase in seizure frequency within 2 weeks prior to enrollment
* Patients 2-17 years of age must have a blood pressure that is =< 95th percentile for age, height, and sex at the time of enrollment. Patients >= 18 years of age must have a blood pressure =< 130/80 mmHg at the time of enrollment (with or without the use of antihypertensive medications).

  * Note: Adequate blood pressure can be achieved using medication for the treatment of hypertension
* All patients must have ophthalmology toxicity assessments performed within 8 weeks prior to enrollment
* For all patients, an MRI of the brain (with orbital cuts for optic pathway tumors) and/or spine (depending on the site(s) of primary disease) with and without contrast must be performed within 8 weeks prior to enrollment
* For patients who undergo a surgery on the target tumor (not required), a pre- and post-operative* MRI of the brain (with orbital cuts for optic pathway tumors) or spine (depending on the site(s) of primary disease) with and without contrast must also be performed. The post-operative MRI must be performed within 4 weeks prior to enrollment. If only a biopsy is performed, a post-operative MRI is not required and the pre-operative (op) MRI within 8 weeks of enrollment will be used as the baseline scan

  * The post-operative MRIs should be performed ideally within 48 hours after surgery if possible
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1, or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Patients must have the ability to swallow whole capsules
* Patients must have receptive and expressive language skills in English, Spanish or French to complete the quality of life (QOL) and neurocognitive assessments
* All patients and/or their parents or legal guardians must sign a written informed consent.
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met.

Exclusion Criteria:

* Patients must not have received any prior tumor-directed therapy including chemotherapy, radiation therapy, immunotherapy, or bone marrow transplant. Prior surgical intervention is permitted
* Patients with a concurrent malignancy or history of treatment (other than surgery) for another tumor within the last year are ineligible
* Patients may not be receiving any other investigational agents
* Patients with any serious medical or psychiatric illness/ condition, including substance use disorders likely in the judgement of the investigator to interfere or limit compliance with study requirements/treatment are not eligible
* Patients who, in the opinion of the investigator, are not able to comply with the study procedures are not eligible
* Female patients who are pregnant are not eligible since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential
* Lactating females who plan to breastfeed their infants are not eligible
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation and for 12 weeks after stopping study therapy are not eligible

  * Note: Women of child-bearing potential and males with sexual partners who are pregnant or who could become pregnant (i.e., women of child-bearing potential) should use effective methods of contraception for the duration of the study and for 12 weeks after stopping study therapy to avoid pregnancy and/or potential adverse effects on the developing embryo
* Cardiac conditions:

  * Known genetic disorder that increases risk for coronary artery disease. Note: The presence of dyslipidemia in a family with a history of myocardial infarction is not in itself an exclusion unless there is a known genetic disorder documented
  * Symptomatic heart failure
  * New York Heart Association (NYHA) class II-IV prior or current cardiomyopathy
  * Severe valvular heart disease
  * History of atrial fibrillation
* Ophthalmologic conditions:

  * Current or past history of central serous retinopathy
  * Current or past history of retinal vein occlusion or retinal detachment
  * Patients with uncontrolled glaucoma

    * If checking pressure is clinically indicated, patients with intraocular pressure (IOP) > 22 mmHg or ULN adjusted by age are not eligible
  * Ophthalmological findings secondary to long-standing optic pathway glioma (such as visual loss, optic nerve pallor, or strabismus) or longstanding orbito-temporal plexiform neurofibroma (PN), such as visual loss, strabismus) will NOT be considered a significant abnormality for the purposes of the study
* Treatments and/or medications patient is receiving that would make her/him ineligible, such as:

  * Supplementation with vitamin E greater than 100% of the daily recommended dose. Any multivitamin containing vitamin E must be stopped prior to study enrollment even if less than 100% of the daily recommended dosing for vitamin E
  * Surgery within 2 weeks prior to enrollment, with the exception of surgical placement for vascular access or cerebrospinal fluid (CSF) diverting procedures such as endoscopic third ventriculostomy (ETV) and ventriculo-peritoneal (VP) shunt.

    * Note: Patients must have healed from any prior surgery prior to enrollment
* Patients who have an uncontrolled infection are not eligible

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 165 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | From randomization to the first occurrence of any of the following events: clinical or radiographic disease progression, disease recurrence, second malignant neoplasm, or death from any cause, assessed up to 3 years after accrual completion
  EFS is defined as time from randomization to the first occurrence of any of the following events: clinical or radiographic disease progression, disease recurrence, second malignant neoplasm, or death from any cause. Patients who are event-free will be censored at the time of last follow-up. Will estimate the hazard ratio based on a stratified Cox proportional hazards model and use Kaplan Meier (KM) methods to visualize and summarize the data.
Number of participants with visual acuity (VA) improvement per arm | Baseline and end of about 12 months of treatment
  VA will be assessed using Teller acuity cards (TAC). A significant improvement in VA will be defined as a decrease of >= 0.2 logMAR (corrected for age) from baseline (pre-treatment baseline) to end of about 12 months of treatment. The primary analysis will be based on per subject outcome (rather than per eye).

SECONDARY OUTCOMES:
Radiographic tumor response rate | Assessed up to 3 years after accrual completion
  Tumors will be classified into complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD). Radiologic response rates will be summarized per arm and be tested for a difference between the two arms using an exact binomial test.
Overall survival (OS) | From randomization until death from any cause or till the time of last follow-up for patients who are alive at the time of analysis, assessed up to 3 years after accrual completion
  OS is defined as the time from randomization until death from any cause or till the time of last follow-up for patients who are alive at the time of analysis. Will use the KM methods, log-rank tests, and Cox proportional hazards models to determine whether there is a difference in OS between the two arms.
Change in VA using HOTV letter acuity testing | Baseline and end of about 12 months of treatment
  HOTV is a recognition acuity measure. It will be conducted on patients who are developmentally able to perform this testing.
Change in motor function | Baseline and approximately 12 months of treatment
  The Vineland-3 Motor Scale from the Comprehensive Parent Rating Form will be used to assess motor deficits. Change in Vineland motor scale from baseline to about 12 months of treatment will be compared between two treatment arms.
Change in quality of life (QOL) | Baseline and 12 months of treatment
  Will be measured by Pain and Hurt subscale score. QOL will be assessed by Pediatric Quality of Life (PedsQL) Generic and Brain Tumor modules. Analysis will be based on a 2-sample t-test comparing change in Pain and Hurt subscale score from baseline to 12 months for the two arms.
Change in quality of life (QOL) | Baseline and 12 months of treatment
  Will be measured by Movement and Balance subscale score. QOL will be assessed by Pediatric Quality of Life (PedsQL) Generic and Brain Tumor modules. Analysis will be based on a 2-sample t-test comparing change in Movement and Balance subscale score from baseline to 12 months for the two arms.
Change in executive function | Baseline and 24 months of treatment
  Will be measured by BRIEF Cognitive Regulation Index (CRI). Executive function will be measured by age-appropriate Behavior Rating Inventory of Executive Function (BRIEF) questionnaire. Analysis will be based on a 2-sample t-test comparing change in the designated score from baseline to 24 months for the two arms.
Change in neurocognitive function | Baseline and 24 months of treatment
  Will be measured by Cogstate composite score. Neurocognitive function will be measured by a computerized battery (Cogstate) testing. Analysis will be based on a 2-sample t-test comparing change in Cogstate composite score from baseline to 24 months for the two arms.

OTHER OUTCOMES:
Change in circumpapillary retinal nerve fiber layer (cpRNFL) thickness by treatment arm | Baseline and 12 months
  cpRNFL thickness is a measure of optical coherence tomography (OCT). This assessment will be conducted in a subgroup of consenting patients with optic pathway gliomas (OPGs) treated at select COG institutions with the expertise to utilize this technology. Analysis will be conducted on a per-eye basis.
cpRNFL thickness at baseline by visual acuity (VA) treatment response | Baseline and 12 months
  Data will be analyzed on a per-eye basis. Children with OPGs will be classified into decline in VA versus (vs.) stable/improved VA, depending on VA treatment response at 12 months. cpRNFL thickness prior to treatment initiation will be compared.
cpRNFL thickness change over time by visual acuity (VA) treatment response | Baseline and 12 months
  Data will be analyzed on a per-eye basis. Children with OPGs will be classified into decline in VA vs. stable/improved VA, depending on VA treatment response at 12 months. cpRNFL thickness change over time will be compared.
Change in macular ganglion cell - inner plexiform layer (GCIPL) thickness by treatment arm | Baseline and 12 months
  GCIPL thickness is another measure of optical coherence tomography (OCT). This assessment will be conducted in a subgroup of consenting patients with optic pathway gliomas (OPGs) treated at select COG institutions with the expertise to utilize this technology. Analysis will be conducted on a per-eye basis.
GCIPL thickness at baseline by visual acuity (VA) treatment response | Baseline and 12 months
  Data will be analyzed on a per-eye basis. Children with OPGs will be classified into decline in VA vs. stable/improved VA, depending on VA treatment response at 12 months. GCIPL thickness prior to treatment initiation will be compared.
GCIPL thickness change over time by visual acuity (VA) treatment response | Baseline and 12 months
  Data will be analyzed on a per-eye basis. Children with OPGs will be classified into decline in VA vs. stable/improved VA, depending on VA treatment response at 12 months. GCIPL thickness change over time will be compared.
Novel semi-automated volumetric magnetic resonance imaging (MRI) measure at 3 months | 3 months on study
  Optic pathway tumors will be classified into progressive disease (PD), stable disease (SD), partial response (PR), and complete response (CR) using novel semi-automated volumetric MRI measurements. This assessment will include patients with OPGs consenting to volumetric MRI study.
Percent change in tumor size between volumetric measure and traditional 2-dimentional (2-D) measure at 3 months | 3 months on study
  This assessment includes participants with OPGs consenting to volumetric MRI study.
Novel semi-automated volumetric MRI measure at 6 months | 6 months on study
  Optic pathway tumors will be classified into progressive disease (PD), stable disease (SD), partial response (PR), and complete response (CR) using novel semi-automated volumetric MRI measurements. This assessment will include patients with OPGs consenting to volumetric MRI study.
Percent change in tumor size between volumetric measure and traditional 2-dimentional (2-D) measure at 6 months | 6 months on study
  This assessment includes participants with OPGs consenting to volumetric MRI study.
Novel semi-automated volumetric MRI measure at 9 months | 9 months on study
  Optic pathway tumors will be classified into progressive disease (PD), stable disease (SD), partial response (PR), and complete response (CR) using novel semi-automated volumetric MRI measurements. This assessment will include patients with OPGs consenting to volumetric MRI study.
Percent change in tumor size between volumetric measure and traditional 2-dimentional (2-D) measure at 9 months | 9 months on study
  This assessment includes participants with OPGs consenting to volumetric MRI study.
Novel semi-automated volumetric MRI measure at 12 months | 12 months on study
  Optic pathway tumors will be classified into progressive disease (PD), stable disease (SD), partial response (PR), and complete response (CR) using novel semi-automated volumetric MRI measurements. This assessment will include patients with OPGs consenting to volumetric MRI study.
Percent change in tumor size between volumetric measure and traditional 2-dimentional (2-D) measure at 12 months | 12 months on study
  This assessment includes participants with OPGs consenting to volumetric MRI study.
Novel semi-automated volumetric MRI measure at 15 months | 15 months on study
  Optic pathway tumors will be classified into progressive disease (PD), stable disease (SD), partial response (PR), and complete response (CR) using novel semi-automated volumetric MRI measurements. This assessment will include patients with OPGs consenting to volumetric MRI study.
Percent change in tumor size between volumetric measure and traditional 2-dimentional (2-D) measure at 15 months | 15 months on study
  This assessment includes participants with OPGs consenting to volumetric MRI study.
Tumor and blood banking | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason R Fangusaro, Principal Investigator — Children's Oncology Group
Locations (132):
- United States (125):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Banner Children's at Desert, Mesa, Arizona
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Corewell Health Children's, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri Children's Hospital, Columbia, Missouri
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Presbyterian Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - New York Medical College, Valhalla, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - UMC Cancer Center / UMC Health System, Lubbock, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (6):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
- HIMA San Pablo Oncologic Hospital, Caguas, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Bergqvist C, Wolkenstein P. MEK inhibitors in RASopathies. Curr Opin Oncol. 2021 Mar 1;33(2):110-119. doi: 10.1097/CCO.0000000000000711. PMID 33395032